CLINICAL TRIAL: NCT01343238
Title: Short- and Longterm Effects of Physical Activity and Dietary Restriction Postpartum on Women's Weight and Body Composition: a Randomized Study
Brief Title: Short- and Longterm Effects of Physical Activity and Dietary Restriction Postpartum
Acronym: LEVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: K2009-70X-21091-01-3; FAS Dnr: 2006-0339 (Other Grant/Funding Number: Swedish Council for Working Life and Social Research)
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
Keywords: obesity; diet; exercise
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diet (Experimental): 12 week diet modification intervention by dietician
  Interventions: Behavioral: Diet
- Exercise (Experimental): 12 week physical exercise modification intervention by physical therapist
  Interventions: Behavioral: Exercise
- Diet and Exercise (Experimental): 12 week diet and exercise behavioral modification by dietician and physical therapist
  Interventions: Behavioral: Diet and Exercise
- Control (No Intervention): Standard procedure

INTERVENTIONS:
Behavioral: Diet — 12 week diet behavior modification
  Arms: Diet
Behavioral: Exercise — 12 week exercise behavioral intervention
  Arms: Exercise
Behavioral: Diet and Exercise — 12 week diet and exercise behavioral modification intervention
  Arms: Diet and Exercise

SUMMARY:
The study will investigate whether physical exercise, or dietary restrictions, or a combination of both, among overweight and obese postpartum women lead to a significantly larger reduction in weight in a longer perspective, compared to similar women not receiving the intervention. The study also will investigate the effects on body composition, cardiovascular fitness, blood lipids, insulin levels and inflammation markers. In total, 68 women with pre-pregnancy BMI 25 - 34.9 will be randomized at 10 wk postpartum into: (1) physical exercise, (2) dietary restrictions, (3) physical exercise + dietary restrictions and (4) control group. The intervention lasts for 12 wk and longterm effects are measured 1 yr after trial initiation. To date only studies showing short term (12 wk) effects exist. Our study is the first to include four intervention groups, so that separate effects of physical activity and dietary restriction and their interaction, can be assessed. Further, the investigators will estimate effects on body composition taking body water into account and estimate total energy expenditure with higher precision than previously. Overweight and obesity is an escalating problem in Sweden. Sustainable weight reduction programs are urgently needed. During the postpartum period, women may be motivated to lose weight. Information aimed at promoting life style changes among overweight and obese women could in a longer perspective be integrated in the regular maternal health care in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* prepregnant BMI 25-35
* non smoking, single term birth
* intention to breastfeed exclusively for 6 mo

Exclusion Criteria:

* Diseases or medication in mother or child

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-05; Primary Completion 2010-08 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Body weight | 12 weeks
  Weight loss after 12 weeks intervention

SECONDARY OUTCOMES:
body composition | 12 weeks
  Change in body composition after 12 weeks intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anna Winkvist, PhD, Principal Investigator — The Unviersity of Gothenburg
Locations (1):
- The University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Derived] Brekke HK, Bertz F, Rasmussen KM, Bosaeus I, Ellegard L, Winkvist A. Diet and exercise interventions among overweight and obese lactating women: randomized trial of effects on cardiovascular risk factors. PLoS One. 2014 Feb 7;9(2):e88250. doi: 10.1371/journal.pone.0088250. eCollection 2014. PMID 24516621
- [Derived] Hagberg LA, Brekke HK, Bertz F, Winkvist A. Cost-utility analysis of a randomized controlled weight loss trial among lactating overweight/obese women. BMC Public Health. 2014 Jan 15;14:38. doi: 10.1186/1471-2458-14-38. PMID 24428802
- [Derived] Winkvist A, Bertz F, Ellegard L, Bosaeus I, Brekke HK. Metabolic risk profile among overweight and obese lactating women in Sweden. PLoS One. 2013 May 7;8(5):e63629. doi: 10.1371/journal.pone.0063629. Print 2013. PMID 23667649
- [Derived] Bertz F, Brekke HK, Ellegard L, Rasmussen KM, Wennergren M, Winkvist A. Diet and exercise weight-loss trial in lactating overweight and obese women. Am J Clin Nutr. 2012 Oct;96(4):698-705. doi: 10.3945/ajcn.112.040196. Epub 2012 Sep 5. PMID 22952179